CLINICAL TRIAL: NCT06096480
Title: Effect of Bilateral Spinae Erector Block (ESP) and Perioperative Gabapentin on Recovery and Length of Stay in Adolescent Spinal Fusion Patients: A Retrospective Cohort Stud
Brief Title: Effect of Spinae Erector Block (ESP) and Gabapentin on Recovery and Length of Stay in Adolescent Spinal Fusion Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, DELFINA SANCHEZ NOVAS, Anesthesiologist, Hospital Italiano de Buenos Aires
Other Study IDs: 6841
Record Dates: First submitted 2023-10-15; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Adolescent Idiopathic Scoliosis
MeSH Terms: interventions — Gabapentin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MMA group: adolescent spinal fusion patients who received intravenous multimodal analgesic strategy alone
- MMA-ESP-G group: adolescent spinal fusion patients who received a multimodal analgesic strategy in combination with a preoperative ESP block and oral gabapentin
  Interventions: Procedure: gabapentin + bilateral spine erector block

INTERVENTIONS:
Procedure: gabapentin + bilateral spine erector block — preoperative, ultrasound-guided, bilateral ESP block (administration of a local anesthetic mixture of ropivacaine 0.375% and lidocaine 1%) and a 100mg dose of oral gabapentin 4 nights daily before surgery and 2 weeks postoperatively.
  Groups: MMA-ESP-G group

SUMMARY:
A retrospective cohort study comparing time to ambulation (hours) between two groups of adolescent spinal fusion patients: a group who received intravenous multimodal analgesic strategy alone (MMA group) and another group who received a multimodal analgesic strategy in combination with a preoperative ESP block and oral gabapentin (MMA-ESP-G group).

DETAILED DESCRIPTION:
One of the major challenges in postoperative care following posterior spinal fusion (PSF) for adolescent idiopathic scoliosis (AIS) is achieving adequate pain control. Opioid-sparing multimodal anesthetic strategies are crucial for achieving effective postoperative pain control and facilitating early mobilization. The erector spinae (ESP) block has been reported as part of various opioid-sparing strategies for spine surgery. Perioperative oral gabapentin (in different dosing protocols) may contribute to reduce postoperative pain and opioid consumption.

The primary aim of this retrospective study was to compare time to ambulation (hours) between two groups of adolescent spinal fusion patients: a group who received intravenous multimodal analgesic strategy alone (MMA group) and another group who received a multimodal analgesic strategy in combination with a preoperative ESP block and oral gabapentin (MMA-ESP-G group). The secondary aim was to compare intensive care length of stay, perioperative opioid requirements and time to urinary catheter removal between groups.

This is a retrospective review of 34 consecutive adolescent spinal fusion patients during August-September 2023 at Hospital Italiano de Buenos Aires, Argentina. The investigators compared two groups: 1) MMA group received an intravenous multimodal analgesic strategy, 2) MMA-ESP-G group received an intravenous multimodal analgesic strategy in combination with a preoperative, ultrasound-guided, bilateral ESP block (administration of a local anesthetic mixture of ropivacaine 0.375% and lidocaine 1%) and a 100mg dose of oral gabapentin 4 nights daily before surgery and 2 weeks postoperatively. Both strategies were protocolized at our institution.

Data was analyzed for the primary outcome: median time to ambulation difference between groups. Differences were considered statistically significant at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of adolescent idiopathic scoliosis (AIS) and primary surgical indication between January 2018 and August 2023.
* ASA patients (American Society of Anesthesiology classification) I to III.

Exclusion criteria:

* Patients who, at the end of the procedure, were transferred to the PICU (Pediatric Intensive Care Unit) on mechanical ventilation.
* Patients undergoing corrective scoliosis surgery in combination with any other surgical procedure.
* Patients who received ESP block postoperatively (Group EM-ESP-G).

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: adolescent spinal fusion patients from Hospital Italiano de Buenos Aires
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-12 (Estimated)

PRIMARY OUTCOMES:
time to ambulation | through study completion, an average of 6 weeks
  time to ambulation (hours)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Italiano de Buenos Aires, Ciudad Autonoma de Buenos Aire, Buenos Aires, Argentina